CLINICAL TRIAL: NCT05458908
Title: ProSPective Evaluation of the dIagnostic Accuracy of siNe spiN Noncontrast Flat-dEtectoR CT (FDCT) for the Detection of Intracranial Hemorrhage in Stroke Patients
Brief Title: ProSPective Evaluation of Non-contrast sINe spiN Flat-dEtectoR CT for the Detection of Intracranial hemorrhageS
Acronym: SPINNERS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Siemens Healthineers AG (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: qu20Psychogios_SPINNERS
Record Dates: First submitted 2022-06-20; First posted 2022-07-14 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Stroke
Keywords: hemorrhagic stroke; ischemic stroke; large-vessel occlusions (LVO); cone beam CT; intracranial hemorrhage; flat detector computer tomography (FDCT)
MeSH Terms: conditions — Stroke; Hemorrhagic Stroke; Ischemic Stroke; Intracranial Hemorrhages

STUDY DESIGN:
Intervention Model Description: Cross-sectional non-inferiority investigation with prospective open label data collection and blinded endpoint assessment
Masking Description: Blinded assessment of outcome events through an independent Core-Lab
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cranial non-contrast syngo DynaCT Sine Spin scan (Experimental): There is only one arm as all patients undergo the same intervention. Subjects with clinical features/symptoms of a stroke (hemorrhagic and non-hemorrhagic stroke patients) will be enrolled. All patients will undergo first a non-contrast MDCT scan and then a non-contrast syngo DynaCT Sine Spin head scan within a maximum timespan of 4 hours between both scans. Only patients in which no invasive procedure in between is planned can be enrolled.
  Interventions: Diagnostic Test: Non-contrast cranial MDCT head scan; Diagnostic Test: Non-contrast syngo DynaCT Sine Spin head scan and application software

INTERVENTIONS:
Diagnostic Test: Non-contrast cranial MDCT head scan — Non-contrast cranial MDCT imaging for visualization of the brain parenchyma (the choice of the device is up to the investigator)
Diagnostic Test: Non-contrast syngo DynaCT Sine Spin head scan and application software — Non-contrast syngo DynaCT Sine Spin imaging for visualization of the brain parenchyma with ARTIS icono biplane angiography system and syngo application software with syngo DynaCT Sine Spin 3-D head imaging protocol.

SUMMARY:
Stroke is one of the leading causes of mortality and disability worldwide. Optimization of intra-hospital pathways is as of today one of the most promising research topics in stroke treatment. A potential solution to shorten the time needed for current workflows, and therefore reperfusion, is to do both imaging and subsequent endovascular therapy (EVT) in the angiography suite using non-contrast syngo DynaCT Sine Spin (FDCT) for the exclusion of intracranial hemorrhage and flat detector CT angiography (FDCTA) or digital subtraction angiography for diagnosis of LVO. It is still a matter of debate if FDCT can reliably differentiate between ischemic and hemorrhagic stroke.

This study aims to investigate if non-contrast syngo DynaCT Sine Spin imaging is non-inferior to non-contrast MDCT imaging regarding its sensitivity and specificity for the detection of intracranial hemorrhages.

DETAILED DESCRIPTION:
Despite concerted efforts, stroke is still one of the leading causes of mortality and disability worldwide.Stroke can be divided into two main types: ischemic and hemorrhagic stroke. Endovascular therapy (EVT) became the gold-standard for the treatment of acute ischemic stroke due to large-vessel occlusions (LVO). However, as was shown by a post-hoc meta-analysis of five trials clinical outcome is highly associated with the time from hospital admission to treatment.

One possibility to substantially shorten this time span is the implementation of a One Stop Management approach. In this workflow both imaging and subsequent EVT is done in the angiography suite using non-contrast flat detector CT (FDCT) for the exclusion of an intracranial hemorrhage. Such workflows dramatically reduce intra-hospital time delays (median reductions of more than 30 minutes) and are associated with improved patient outcomes. One of the biggest hurdles for a large-scale implementation of a One Stop Management approach up to now is the ability to differentiate between ischemic and hemorrhagic stroke with FDCT. In a recent study we have reported very high sensitivity and specificity for the detection of intracranial hemorrhage with FDCT.

Recently Siemens Healthineers introduced the new ARTIS icono angiography system with a new non-contrast syngo DynaCT Sine Spin protocol FDCT, which should improve the quality and soft tissue resolution of native cranial FDCT scans especially in the posterior fossa and skull base. Therefore, the study aims to evaluate if non-contrast syngo DynaCT Sine Spin FDCT is non-inferior to non-contrast multidetector CT (MDCT) for the detection of intracranial hemorrhages.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent as documented by signature or fulfilling the criteria for emergency or deferral consent
* Patients with symptoms suggestive of ischemic stroke (NIHSS ≥ 7) or suggestive of haemorrhagic stroke with a cranial non-contrast MDCT and a feasible non-contrast syngo DynaCT Sine Spin within 4 hours
* Patient presenting within 24 hours of last seen well
* Patients presenting directly to the treating hospital (i.e. mothership patients) OR transfer patients with the indication for repeated imaging according to the standard operation procedures of the treating hospital
* Age above 18 years
* Agreement of treating physician to perform non-contrast syngo DynaCT Sine Spin

Exclusion Criteria:

* Severe metal artifacts on initial MDCT imaging
* Planned invasive interventions between MDCT and FDCT scan
* Clinical deterioration between MDCT and FDCT scan (i.e. an increase of the NIHSS of more than 4 points)
* Evidence of an ongoing pregnancy prior to enrollment. A negative pregnancy test before enrollment is required for all women with child-bearing potential

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Estimated)
Dates: Start 2022-10-25 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Occurrence of an intracranial hemorrhage (yes/no) | Day 0 - within 4 hours of enrollment
  The primary outcome is the occurrence of intracranial hemorrhages (yes vs no) as assessed by a blinded core-lab. The primary outcome will be used to calculate the sensitivity and specificity of non-contrast syngo DynaCT Sine Spin imaging for the detection of intracranial hemorrhages.
  The primary outcome will be assessed on both scans.

OTHER OUTCOMES:
Change in Adverse Device Events (ADEs) | At 24 h ± 6h after enrollment
  All device related adverse events (ADEs) will be evaluated up to 24 hours after the study intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Marios-Nikos Psychogios, Prof Dr, Principal Investigator — University Hospital, Basel, Switzerland; Nitin Goyal, MD, Study Chair — Semmes Murphey Clinic and University of Tennessee Health Sciences Center
Locations (14):
- United States (8):
  - Swedish Medical Center, Denver, Colorado
  - AdvocateAurora Health, Chicago, Illinois
  - Nortshore University Health System, Chicago, Illinois
  - New York University Langone Health, New York, New York
  - Mount Sinai Health System, New York, New York
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Semmes Murphy Clinic, Memphis, Tennessee
  - University of Virginia Health System, Charlottesville, Virginia
- HUS, Helsinki, Helsinki, Finland
- CHRU de Tours, Tours, France
- Hospital Vall d'Hebron, Barcelona, Barcelona, Spain
- Switzerland (3):
  - University Hospital Basel, Basel
  - Inselspital Bern, Bern
  - Kantonsspital Luzern, Lucerne

REFERENCES:
- [Background] Meier T, Dimroth P. Intersubunit bridging by Na+ ions as a rationale for the unusual stability of the c-rings of Na+-translocating F1F0 ATP synthases. EMBO Rep. 2002 Nov;3(11):1094-8. doi: 10.1093/embo-reports/kvf216. Epub 2002 Oct 22. PMID 12393753
- [Background] Petroulia VD, Kaesmacher J, Piechowiak EI, Dobrocky T, Pilgram-Pastor SM, Gralla J, Wagner F, Mordasini P. Evaluation of Sine Spin flat detector CT imaging compared with multidetector CT. J Neurointerv Surg. 2023 Mar;15(3):292-297. doi: 10.1136/neurintsurg-2021-018312. Epub 2022 Mar 22. PMID 35318960
- [Background] Psychogios MN, Behme D, Schregel K, Tsogkas I, Maier IL, Leyhe JR, Zapf A, Tran J, Bahr M, Liman J, Knauth M. One-Stop Management of Acute Stroke Patients: Minimizing Door-to-Reperfusion Times. Stroke. 2017 Nov;48(11):3152-3155. doi: 10.1161/STROKEAHA.117.018077. Epub 2017 Oct 10. PMID 29018132
- [Background] Leyhe JR, Tsogkas I, Hesse AC, Behme D, Schregel K, Papageorgiou I, Liman J, Knauth M, Psychogios MN. Latest generation of flat detector CT as a peri-interventional diagnostic tool: a comparative study with multidetector CT. J Neurointerv Surg. 2017 Dec;9(12):1253-1257. doi: 10.1136/neurintsurg-2016-012866. Epub 2016 Dec 20. PMID 27998955
- [Derived] Psychogios M, Brehm A, Goyal N, Boulouis G, Burkhardt JK, Chowdhry SA, Frei D, Gralla J, Kaesmacher J, Kellogg RT, Kellner CP, Lopes DK, Raz E, Strbian D, Mannismaki L, Tomasello A, Tsogkas I, von Hessling A, Karwacki GM, Guzman R, Rommers N, Liebeskind DS, Arthur AS; SPINNERS investigators. ProSPective evaluation of the dIagnostic accuracy of siNe spiN non-contrast flatdEtectoR CT (FDCT) for the detection of intracranial hemorrhage in stroke patients - Protocol of a non-inferiority comparison to multi detector CT. PLoS One. 2025 Aug 28;20(8):e0330608. doi: 10.1371/journal.pone.0330608. eCollection 2025. PMID 40875663